CLINICAL TRIAL: NCT07050784
Title: A Crossover Randomized Controlled Trial Comparing Smart Textile and Hydrogel Electrodes for Neurostimulation in Healthy Adults
Brief Title: Wearable Garment vs Gel Electrodes for Electrical Muscle Stimulation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Myant Medical Corp. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 157491
Record Dates: First submitted 2025-06-09; First posted 2025-07-03 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Healthy
Keywords: Textile electrodes; Smart clothing; Neuromuscular electrical stimulation; Transcutaneous electrical nerve stimulation; Functional electrical stimulation

STUDY DESIGN:
Intervention Model Description: Crossover randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Hydrogel electrodes (Active Comparator): Gold-standard comparator
  Interventions: Device: Hydrogel electrodes
- Dry polymer-textile electrodes with Skin Lotion A (Experimental)
  Interventions: Device: Dry polymer-textile electrodes with Skin Lotion A
- Dry textile electrodes with gel pads attached to the electrode (Experimental)
  Interventions: Device: Dry textile electrodes with gel pads attached to the electrode
- Dry polymer-textile electrodes with Skin Lotion B (Experimental)
  Interventions: Device: Dry polymer-textile electrodes with Skin Lotion B
- Dry polymer-textile electrodes with Skin Lotion C (Experimental)
  Interventions: Device: Dry polymer-textile electrodes with Skin Lotion C

INTERVENTIONS:
Device: Hydrogel electrodes — Neurostimulation using standard self-adhesive hydrogel electrodes
  Arms: Hydrogel electrodes
Device: Dry polymer-textile electrodes with Skin Lotion A — Neurostimulation with dry polymer-textile electrodes using Skin Lotion A
  Arms: Dry polymer-textile electrodes with Skin Lotion A
Device: Dry textile electrodes with gel pads attached to the electrode — Neurostimulation with dry textile electrodes with gel pads attached to the electrode
  Arms: Dry textile electrodes with gel pads attached to the electrode
Device: Dry polymer-textile electrodes with Skin Lotion B — Neurostimulation with dry polymer-textile electrodes with Skin Lotion B
  Arms: Dry polymer-textile electrodes with Skin Lotion B
Device: Dry polymer-textile electrodes with Skin Lotion C — Neurostimulation with dry polymer-textile electrodes using Skin Lotion C
  Arms: Dry polymer-textile electrodes with Skin Lotion C

SUMMARY:
The goal of this study is to evaluate whether textile-based electrodes can provide neurostimulation that is comparable in comfort and effectiveness to traditional hydrogel electrodes in healthy adults.

The main questions it aims to answer are:

1. Is the perceived sensation of stimulation using textile electrodes non-inferior to that of hydrogel electrodes?
2. Is the current required to evoke muscle contractions similar between textile and hydrogel electrodes?

Each participant will complete three stimulation conditions in random order across separate visits:

1. hydrogel electrodes (standard),
2. dry polymer-textile electrodes with lotion, and
3. dry textile electrodes with hydrogel pads

Electrical stimulation will be delivered to the lower leg muscles using a wearable sleeve with integrated electrodes. The investigators will assess sensorimotor thresholds (e.g., detection, motor, and full motor threshold), skin-electrode impedance, and torque. Participants will also rate stimulation comfort, intensity, and sensation location via questionnaire.

After the three primary arms, participants may optionally complete two additional arms using different moisturizers applied to the textile electrodes to evaluate their impact on stimulation performance.

The results of this study will help determine whether textile electrodes can be used as an effective and comfortable alternative to hydrogel electrodes in wearable neurostimulation applications.

DETAILED DESCRIPTION:
Neurostimulation involves the use of electric current delivered through skin-surface electrodes to activate muscles. It is commonly used for purposes such as muscle strengthening, motor function improvement, blood flow enhancement, and in neuroprostheses. Standard neurostimulation systems typically rely on disposable hydrogel electrodes, which can cause skin irritation and tend to dry out over time. These limitations make hydrogel electrodes less suitable for long-term or repeated use.

Textile-based electrodes are an emerging alternative. These electrodes are integrated into wearable garments, making them washable, reusable, and more comfortable for extended wear times. However, research directly comparing their effectiveness and user experience compared to hydrogel electrodes is limited.

The goal of this study is to compare textile electrodes to gold-standard hydrogel electrodes for muscle activation and perceived stimulation sensation. The investigators hypothesize that: 1) there will be no clinically meaningful difference in participants' perception of the stimulation between textile and hydrogel electrodes, and 2) there will be no significant difference in the stimulation current required to elicit functional contractions.

This is a crossover randomized controlled trial involving three primary arms: 1) hydrogel electrodes, 2) dry polymer-textile electrodes with lotion, and 3) dry textile electrodes with gel pads applied. Each participant will perform all three arms in a randomized order with at least 24 hours between visits. Stimulation will be delivered to the calf and tibialis anterior muscles using the same electrical stimulator and settings in all conditions. Following completion of the three primary arms, participants will be given the option to complete an additional two arms using different types of commercially available moisturizers on the dry textile electrodes to assess comparative on-body performance of different water-based moisturizers. All moisturizers are commercially available and are labelled Skin Lotion A, B, and C in the 'Arms and Interventions' section.

A sample size of 18 participants is required to detect a Cohen's f of 0.40 with 95% power and a significance level of ⍺ = 0.05 for a within-subjects one-way repeated measures analysis of variance (ANOVA) with three conditions. To preserve statistical power, the investigators will recruit 20 participants. Pilot data comparing textile to hydrogel electrodes provided an estimated effect size of f = 0.65. Given the pilot data was not randomized, which likely inflated the observed effect size, the investigators conservatively based their sample size calculation on a Cohen's f of 0.40 (i.e., a large effect size) to ensure adequate power to detect a potentially smaller true effect.

A non-inferiority analysis will compare perceived stimulation intensity on a 10-point numerical rating scale. A 2-point difference is set as the non-inferiority margin based on prior research on the minimal clinically important difference. Textile electrodes will be considered non-inferior if the upper bound of the 95% confidence interval for the difference in intensity remains below this threshold. Repeated measures ANOVAs and Tukey's post hoc tests will be used to analyze the outcome variables where appropriate.

ELIGIBILITY:
Inclusion Criteria:

* Healthy (without a known diagnosis of cardiovascular, pulmonary or neurological condition)

Exclusion Criteria:

* Known pregnancy
* Implanted defibrillator or pacemaker
* Pain in the body part being tested
* Open wound or dressing (e.g. band-aid) on a body part that needs to be in contact with the electrodes
* Severe frailty such that donning or doffing the garment may cause a danger of falling

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Perceived intensity of stimulation | At each of the 5 study visits (Visit 1 through Visit 5) over approximately a 3-week period.
  Participants will rate the perceived intensity of electrical stimulation at the current required to elicit 20% of their maximal voluntary contraction (MVC). Intensity will be assessed using a 10-point numerical scale, where 0 represents no sensation and 10 represents painful stimulation.

SECONDARY OUTCOMES:
Sensorimotor responses to electrical stimulation | At each of the 5 study visits (Visit 1 through Visit 5) over approximately a 3-week period.
  Current amplitude required to elicit various sensorimotor responses will be recorded.
  Participants will receive electrical stimulation to the lower leg. The study will measure:
  * Detection threshold: the smallest current the participant can feel.
  * Motion threshold: the lowest current that causes visible movement.
  * Full range of motion amplitude: the current needed for full joint range of motion.
  * Just noticeable difference: the smallest change in current a participant can detect.
  Stimulation will be increased gradually and stopped if discomfort is reported. All stimulation will not exceed safe current limits (i.e., 100 mA).
Kinematic recruitment curves | At each of the 5 study visits (Visit 1 through Visit 5) over approximately a 3-week period.
  Kinematic recruitment curves will be created by measuring ankle movement during stimulation. A camera will record the ankle as stimulation amplitude increases in small increments. Joint angles will be measured from the video and plotted against stimulation intensity to produce kinematic recruitment curves.
Torque | At each of the 5 study visits (Visit 1 through Visit 5) over approximately a 3-week period.
  Maximum voluntary contraction (MVC) will be determined through three maximal effort contractions of the ankle. Electrical stimulation will then be applied to determine the current required to produce 20% of the MVC.
Sensation questionnaire | At each of the 5 study visits (Visit 1 through Visit 5) over approximately a 3-week period.
  Participants will complete a questionnaire following stimulation to report:
  * How the stimulation felt
  * Where it was felt
  * How comfortable it was, rated on a 7-point scale, with 0 being comfortable and 7 being uncomfortable
Skin-electrode impedance | At each of the 5 study visits (Visit 1 through Visit 5) over approximately a 3-week period.
  To measure electrical impedance, a small electrical signal will be sent through the electrodes across a range of frequencies, and resistance will be recorded. This helps evaluate how well the electrodes conduct current during use.

CONTACTS AND LOCATIONS:
Overall Officials: Milad Alizadeh Meghrazi, Principal Investigator — Myant Medical Corp.
Locations (1):
- Myant Medical Corp, Mississauga, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Study is internal